CLINICAL TRIAL: NCT02275858
Title: A Double Blind, Placebo Controlled, Randomized Cross Over Study of an Enteroscope Stiffening Device to Increase Terminal Ileum Intubation Rate During Retrograde Balloon Assisted Enteroscopy
Brief Title: Enteroscopy Stiffening Device for Retrograde Balloon Assisted Enteroscopy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped due to carry over effect in the cross over study design.
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Michael Sai Lai Sey, MD, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: HSREB#105974
Record Dates: First submitted 2014-10-23; First posted 2014-10-27 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Small Bowel Diseases
Keywords: balloon assisted enteroscopy; terminal ileum intubation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stiffening wire first (Experimental): This arm will use the stiffening wire first followed by the placebo wire
  Interventions: Device: Stiffening wire; Device: Placebo wire
- Placebo wire first (Placebo Comparator): This arm will use the placebo wire first followed by the stiffening wire
  Interventions: Device: Stiffening wire; Device: Placebo wire

INTERVENTIONS:
Device: Stiffening wire — Stiffening wire
Device: Placebo wire — Placebo wire

SUMMARY:
Balloon assisted enteroscopy has revolutionized the management of small bowel diseases by enabling endoscopic access deep into the small bowel. Using a combination of antegrade (through the mouth) and retrograde (through the anus) approaches, a large portion of the small bowel can be examined. Access to the proximal small bowel through the pylorus using the antegrade approach is straightforward but intubating the distal small bowel through the ileocecal valve is challenging due to the flexibility of the enteroscope. Recently, an enteroscopy stiffening wire has been developed. The purpose of our double blind placebo controlled randomized cross over study is to evaluate the performance of the enteroscopy stiffening wire in achieving terminal ileum intubation (TI) during retrograde balloon assisted enteroscopy.

DETAILED DESCRIPTION:
Small bowel endoscopy has undergone a paradigm shift in the past decade. Prior to this, the small bowel was considered a 'black hole' due to our inability to visualize it endoscopically and the limited sensitivity of radiologic studies. This all changed with the development of video capsule endoscopy, which gave physicians the ability to visualize the full length of the small bowel. Although widely considered a great leap forward, video capsule endoscopy is limited by its inability to perform any form of endoscopic intervention. Thus, something was needed to biopsy and treat the diseases detected with video capsule endoscopy. Double balloon enteroscopy (DBE) was invented in Japan in 2001.(1) Using an overtube and two inflatable balloons, DBE enabled deep intubation of the small bowel through a series of push and pull maneuvers to accordion the small bowel over the overtube. This procedure proved highly successful in the diagnosis and treatment of small bowel diseases.(2, 3) Subsequently, single balloon enteroscopy (SBE) was developed consisting of a single overtube balloon.(4, 5) Collectively, these techniques are called balloon assisted enteroscopy.

Balloon assisted enteroscopy can be performed using an antegrade (through the mouth) or retrograde (through the anus) approach. The two approaches are considered complimentary since the antegrade approach enables visualization of the proximal and mid small bowel while the distal portion is seen with the retrograde approach. Of the two, the retrograde approach is more challenging as it requires first going through the length of the colon followed by intubation of the terminal ileum (TI) to reach the small bowel. TI intubation during balloon assisted enteroscopy can be difficult due to the inherent flexibility of the enteroscope.(6) Even in expert hands, the success rate for TI intubation ranges between 69-79% (7-9) and takes on average 28 minutes to intubate once the cecum has been reached.(8) Patients with distal ileum lesions who fail retrograde balloon assisted enteroscopy have limited options and may require surgery.

Recently, an enteroscopy stiffening wire has been developed by Zutron Medical LLC (Kansas, USA). This is a through the scope wire that stiffens the enteroscope to increase the maximal depth of insertion. Since the difficulty in intubating the TI during retrograde balloon assisted enteroscopy is largely due to the inherent flexibility of the enteroscope, a stiffening wire may improve the ease of TI intubation. The objective of our double blind placebo controlled crossover study is to evaluate the performance of the enteroscopy stiffening wire in improving TI intubation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing retrograde balloon assisted enteroscopy (either SBE or DBE) for management of small bowel diseases.

Exclusion Criteria:

1. Age < 14
2. Prior ileocecal surgery, resection, or anastomosis
3. Inability to reach the cecum during retrograde balloon assisted enteroscopy
4. Hemodynamic instability
5. Inpatient procedure

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Terminal ileum intubation rate | Intraoperative

SECONDARY OUTCOMES:
Terminal ileum intubation time for successful intubations | Intraoperative
Small bowel diagnostic rate | Intraoperative
Small bowel intervention rate | Intraoperative

OTHER OUTCOMES:
Peri-procedural adverse events | Within the first 24 hours of the procedure
Adverse events within the first 7 days | Between 1-7 days of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sey, MD, Principal Investigator — London Health Sciences Centre-Victoria Campus
Locations (1):
- London Health Sciences Center-Victoria Campus, London, Ontario, Canada

REFERENCES:
- [Background] Yamamoto H, Sekine Y, Sato Y, Higashizawa T, Miyata T, Iino S, Ido K, Sugano K. Total enteroscopy with a nonsurgical steerable double-balloon method. Gastrointest Endosc. 2001 Feb;53(2):216-20. doi: 10.1067/mge.2001.112181. PMID 11174299
- [Background] Yamamoto H, Kita H, Sunada K, Hayashi Y, Sato H, Yano T, Iwamoto M, Sekine Y, Miyata T, Kuno A, Ajibe H, Ido K, Sugano K. Clinical outcomes of double-balloon endoscopy for the diagnosis and treatment of small-intestinal diseases. Clin Gastroenterol Hepatol. 2004 Nov;2(11):1010-6. doi: 10.1016/s1542-3565(04)00453-7. PMID 15551254
- [Background] May A, Nachbar L, Ell C. Double-balloon enteroscopy (push-and-pull enteroscopy) of the small bowel: feasibility and diagnostic and therapeutic yield in patients with suspected small bowel disease. Gastrointest Endosc. 2005 Jul;62(1):62-70. doi: 10.1016/s0016-5107(05)01586-5. PMID 15990821
- [Background] Hartmann D, Eickhoff A, Tamm R, Riemann JF. Balloon-assisted enteroscopy using a single-balloon technique. Endoscopy. 2007 Feb;39 Suppl 1:E276. doi: 10.1055/s-2007-966616. Epub 2007 Oct 24. No abstract available. PMID 17957636
- [Background] Kawamura T, Yasuda K, Tanaka K, Uno K, Ueda M, Sanada K, Nakajima M. Clinical evaluation of a newly developed single-balloon enteroscope. Gastrointest Endosc. 2008 Dec;68(6):1112-6. doi: 10.1016/j.gie.2008.03.1063. Epub 2008 Jul 2. PMID 18599052
- [Background] ASGE Training Committee 2011-2012; Rajan EA, Pais SA, Degregorio BT, Adler DG, Al-Haddad M, Bakis G, Coyle WJ, Davila RE, Dimaio CJ, Enestvedt BK, Jorgensen J, Lee LS, Mullady DK, Obstein KL, Sedlack RE, Tierney WM, Faulx AL. Small-bowel endoscopy core curriculum. Gastrointest Endosc. 2013 Jan;77(1):1-6. doi: 10.1016/j.gie.2012.09.023. PMID 23261090
- [Background] Mehdizadeh S, Ross A, Gerson L, Leighton J, Chen A, Schembre D, Chen G, Semrad C, Kamal A, Harrison EM, Binmoeller K, Waxman I, Kozarek R, Lo SK. What is the learning curve associated with double-balloon enteroscopy? Technical details and early experience in 6 U.S. tertiary care centers. Gastrointest Endosc. 2006 Nov;64(5):740-50. doi: 10.1016/j.gie.2006.05.022. PMID 17055868
- [Background] Mehdizadeh S, Han NJ, Cheng DW, Chen GC, Lo SK. Success rate of retrograde double-balloon enteroscopy. Gastrointest Endosc. 2007 Apr;65(4):633-9. doi: 10.1016/j.gie.2006.12.038. PMID 17383460
- [Background] Tee HP, How SH, Kaffes AJ. Learning curve for double-balloon enteroscopy: Findings from an analysis of 282 procedures. World J Gastrointest Endosc. 2012 Aug 16;4(8):368-72. doi: 10.4253/wjge.v4.i8.368. PMID 22912911